CLINICAL TRIAL: NCT05685199
Title: Identifying the Determinants of Bleeding and Hypermobility in Patients With Heavy Menstrual Bleeding
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Wallace H. Coulter Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IDBLEED
Record Dates: First submitted 2022-12-15; First posted 2023-01-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hypermobile Ehlers-Danlos Syndrome; Heavy Menstrual Bleeding; Hypermobility Syndrome (Disorder)
Keywords: Heavy Menstrual Bleeding; Joint Hypermobility; Hypermobile Ehlers-Danlos Syndrome; Generalized joint Hypermobility Syndrome Disorder; Loose Joints
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3; Menorrhagia; Joint Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will provide a sample of blood for banking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: Participants with heavy menstrual bleeding (HMB)
- Control Group: Participants without heavy menstrual bleeding (HMB)

SUMMARY:
In this study, researchers want to learn about the connection between heavy bleeding issues and joint hypermobility (loose joints). They want to know if these issues may indicate other connective tissue problems in girls and women with heavy menstrual bleeding who do not have a known cause.

Primary Objective

* Compare the severity of heavy menstrual bleeding (HMB) in women with and without Generalized joint Hypermobility Syndrome Disorder/hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS) using bleeding scores.

Secondary Objectives

* Compare the frequency of co-morbidities in women with and without G-HSD/hEDS.

DETAILED DESCRIPTION:
Patients will be eligible for inclusion and offered to be screened for enrollment in this study if the duration of their menses was greater than or equal to 7 days, and they reported either "flooding" or bleeding through a tampon or napkin in 2 hours or less with most periods, have no identifiable bleeding disorder, and have evidence of severe iron deficiency anemia (hemoglobin < 8 g/dL).

Once enrolled, joint hypermobility will be evaluated using a Beighton score which will be used to assign participants to two groups: with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS). Participants will then undergo a detailed clinical examination to further classify them using the 2017 diagnostic criteria and complete symptom questionnaires. Finally, participants will be consented to TBANK (NCT01354002) and INSIGHT HD (NCT02720679) to provide a sample of leftover blood for banking for future research. Participants will be seen annually for the next 3 years as part of their standard of care to document the course of their symptoms.

Visit 1: Self-BAT Questionnaire, Beighton Score examination, 2017 hEDS examination, PROMIS (Peds/Parent) questionnaire, PHQ15 questionnaire, COMPASS31 questionnaire, Menstrual distress questionnaire (ENDOPAIN), and Heavy menstrual bleeding checklist (both pediatric and adult).

Visit 2: Self-BAT Questionnaire, PROMIS (Peds/Parent) questionnaire, PHQ15 questionnaire, COMPASS31 questionnaire, Menstrual distress questionnaire (ENDOPAIN).

Visit 3: Self-BAT Questionnaire, PROMIS (Peds/Parent) questionnaire, PHQ15 questionnaire, COMPASS31 questionnaire, Menstrual distress questionnaire (ENDOPAIN).

Please note: At the present time patient enrollment is limited to St. Jude established patients only.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 12-40 years
* Presence of HMB
* Evidence of severe iron-deficiency anemia (hemoglobin level of < 8 g/dL)

Exclusion Criteria:

* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Current use of anticoagulant and antiplatelet medications
* Currently pregnant
* Medical conditions that could cause HMB but are not necessarily a bleeding disorder, including, but not limited to:

  * Uncontrolled hypertension
  * Documented uterine structural abnormality
  * Insulin-dependent diabetes mellitus
  * Chronic kidney disease
  * Chronic liver disease
  * Thyroid disease
  * Documented peripheral arterial disease, venous or arterial vascular events in the past
  * A structural pathology that would explain the HMB
* Presence of a bleeding disorder indicated by prothrombin time, activated partial thromboplastin time, fibrinogen, and von Willebrand factor activity, antigen and factor VIII
* Persistent thrombocytopenia as defined by a platelet count of <150,000/uL
* If the participant answers "yes" to any of the following questions, they are ineligible:

  * Could the patient have a known connective tissue disorder?
  * Family history of sudden death
  * Family history/personal history of uterine rupture or bowel perforation
  * Family history/personal history of arterial rupture
  * Family history/personal history of aneurysm
  * Family history/personal history of an established EDS diagnosis based on genetic evaluation

Ages: 12 Years to 40 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — Female
Study Population: Participants who meet the Eligibility criteria and consent
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
Severity of bleeding symptoms in women with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS): Self-Bleeding Assessment Tool (Self-Bat) | Yearly for 3 years
  Summary statistics of bleed score including mean, median, standard deviation and range will be reported for women with and without G-HSD/hEDS. The Self-BAT which consist of 14 categories for assessing bleeding symptom will be used. Each of the 14 variables is scored from 0-4 (except CNS bleeding when the scores are 0, 3 and 4) and on the basis of this a final score is derived. Scores of ≥ 3 in children, ≥ 4 in adult males and ≥ 6 in adult females is considered abnormal.
Number of patients with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS). | Approximately 3 years
  The number of patients with G-HSD/hEDS will be reported
Proportion of patients with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS). | Approximately 3 years
  The proportion of patients with G-HSD/hEDS will be reported

SECONDARY OUTCOMES:
Co-morbidities in women with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS) - PHQ15 | Yearly for 3 years
  Investigators will compare co-morbidities in women with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS) using PHQ 15. The PHQ-15 is a subscale of the full Patient Health Questionnaire (PHQ) and screens for 15 somatic symptoms. It scores symptom presence and severity on a 3-point Likert scale (0-2). The total score ranges from 0-30 with higher values indicating increased severity as follows: Minimal (0-4); Low (5-9); Medium (10-14); High (15-30).
Co-morbidities in women with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS): Peds Patient-reported Outcomes Measurement Information System (PROMIS) 49 and Parent Proxy 49 | Yearly for 3 years
  Investigators will compare co-morbidities in women with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS) using Peds PROMIS 49 and Parent Proxy 49. The Peds PROMIS 49 is self-reported measures of global, physical, mental, and social health for children (ages 8-17) in the general population and those living with a chronic condition. The Parent Proxy 49 is intended for parents serving as proxy for their child (youth ages 5-17). PROMIS scores are reported as T scores ranging from 0-100. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like Anxiety, a T-score of 60 is one SD worse than average. By comparison, an Anxiety T-score of 40 is one SD better than average. However, for positively-worded concepts like Physical Function-Mobility, a T-score of 60 is one SD better than average while a T-score of 40 is one SD worse than average.
Co-morbidities in women with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS): PROMIS 57 | Yearly for 3 years
  Investigators will compare co-morbidities in women with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS) using adult PROMIS 57. The PROMIS 57 is for self-reporting measures of global, physical, mental, and social health for adults in the general population and those living with a chronic condition. PROMIS scores are reported as T scores ranging from 0-100. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like Anxiety, a T-score of 60 is one SD worse than average. By comparison, an Anxiety T-score of 40 is one SD better than average. However, for positively-worded concepts like Physical Function-Mobility, a T-score of 60 is one SD better than average while a T-score of 40 is one SD worse than average.
Co-morbidities in women with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS): Compass 31 | Yearly for 3 years
  Investigators will compare co-morbidities in women with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS) using COMPASS31. The COMPASS31 contains 31 questions with Likert scales ranging in length from 2 to 6 items with higher scores indicating increased severity. COMPASS31 provides raw scores and standardized scores providing a total weighted score (0-100) of severity. The scale yields 6 subscales and a total score as follows: Orthostatic intolerance (4-10), Vasomotor (3-6); Secretomotor (4-7); Gastrointestinal (12-28); Bladder (3-9); Pupillomotor (5-15); Total (31-75)
Co-morbidities in women with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS): Menstrual Distress Questionnaire | Yearly for 3 years
  Investigators will compare co-morbidities in women with and without Generalized joint Hypermobility Syndrome Disorder/ hypermobile Ehlers-Danlos Syndrome (G-HSD/hEDS)using the Menstrual Distress Questionnaire. This is a 21-element survey (ENDOPAIN 4D) which measures the gynecological and pelvic pain symptoms associated with periods. Each question is on a 11-point Likert scale with higher scores reflecting more severe symptoms or symptoms that most closely resemble the description.

CONTACTS AND LOCATIONS:
Overall Officials: Rohith Jesudas, MBBS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols